CLINICAL TRIAL: NCT00179946
Title: Impact of HLA Matching on Outcome in Pediatric Patients Undergoing Unrelated Umbilical Cord Blood Transplantation.
Brief Title: HLA Matching - Unrelated Umbilical Cord Blood Transplantation
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: BMT 0603 HLA
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Histocompatibility Testing

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: HLA typing

SUMMARY:
The aim of this protocol is to clarify the role of HLA matching in unrelated umbilical cord blood (UCB) transplantation and to identify the level of HLA matching required assuring successful outcome of unrelated UCB transplantation.

DETAILED DESCRIPTION:
The aim of this protocol is to clarify the role of HLA matching in unrelated umbilical cord blood (UCB) transplantation and to identify the level of HLA matching required assuring successful outcome of unrelated UCB transplantation.

The study will answer the following questions:

1. Is HLA matching beneficial to unrelated UCB transplantation?
2. Which HLA loci, HLA-A, B, C, DRB1, or BQB1 is/are important to math, or alternatively to mismatch, to improve graft survival?
3. Which HLA loci, HLA-A, B, C, DRB1, or BQB1 mismatches is/are "permissive mismatches" or well tolerated mismatches?
4. What level of typing resolution (low, intermediate, or hgh) is required to perform patient/donor H:A matching?

By studying the cells and blood of donors and recipients, we may learn more about improving the tissue matching between unrelated donors and their recipients. Also, we hope to learn if an additional level of matching testing improves the results of the transplant treatment. Increasing knowledge about tissue matching could result in the improved long-term survival of cord blood transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients undergoing an unrelated umbilical cord blood transplantation.

Exclusion Criteria:

* Refusal to participate in study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Chadhury, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States